CLINICAL TRIAL: NCT03149341
Title: MR Imaging and Computational Simulation of Cardiovascular Physiology Including Velocity, Pressure, and Wall Shear Stress
Brief Title: MRI and Computational Simulation Cardiology Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jeffrey A. Feinstein, MD, MPH. Associate Professor, Pediatrics and, by courtesy, BioEngineering. Director, Pediatric Cardiology Fellowship Program. Director, Vera Moulton Wall Center for Pulmonary Vascular Disease, Stanford University
Other Study IDs: SQL 80004
Record Dates: First submitted 2014-05-13; First posted 2017-05-11 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Congenital Heart Disease; Pulmonary Hypertension
MeSH Terms: conditions — Heart Defects, Congenital; Hypertension, Pulmonary | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study: Congenital heart disease or acquired cardiopulmonary disease who will get (or have gotten) and MRI
  Interventions: Other: Magnetic Resonance Imaging
- Normal Volunteers: No congenital heart disease or acquired cardiopulmonary disease who will get (or have gotten) and MRI
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging — All subjects will undergo or have already undergone Magnetic Resonance Imaging. Normal volunteers will be used for comparison with subjects. To minimize risk, normal volunteers will NOT undergo anesthesia, sedation or receive intravenous contrast during procedure.

SUMMARY:
The purpose of this study is to (1) quantify cardiovascular anatomy and physiology using magnetic resonance imaging under both resting and exercise conditions in patients who have congenital heart disease and in age-matched normal volunteers, (2) use computer models to reproduce and simulate blood flow in these patients, and then (3) to combine the imaging data and computer models to estimate values which cannot be directly measured and to predict physiological changes induced by exercise and medical or surgical therapies.

DETAILED DESCRIPTION:
Investigators hope to gain a greater understanding of the hemodynamics of congenital heart disease and their associated operations as they pertain to real-life situations (i.e. upright and non-sedentary, rest and exercise). With this knowledge, investigators would look to optimize the geometry and physiology of the patients, potentially reducing several of the long-term complications found in congenital heart disease patients such as cardiomyopathy, pulmonary hypertension, arrhythmias, thrombosis and heart failure.

ELIGIBILITY:
Inclusion Criteria:

* patients will have congenital heart disease or acquired cardiopulmonary disease.
* normal volunteers will be willing to undergo MRI

Exclusion Criteria:

* patients unable to receive intravenous contrast material (this does not apply to normal volunteers)
* subjects with arrhythmias which will prevent MRI cardiac gating
* subjects with illnesses which make participation inappropriate. In addition, patients who would normally be excluded from an MRI study because of pacemaker implant, aneurysm clip, severe claustrophobia, or any other condition which, based on the Investigator's judgment, would preclude proximity to a strong magnetic field will be excluded from this study as well.
* NORMAL VOLUNTEERS may be excluded if they are not able to remain still during the exam or follow the instructions of the investigators.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: LPCH and Stanford clinics
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2008-02; Primary Completion 2029-01 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Wall Shear Stress | 20 years
  Computational parameters derived from clinical diagnostic modalities

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Feinstein, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital at Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication